CLINICAL TRIAL: NCT05937399
Title: Project PLUS- Promoting Lung Cancer Screening Among Screening-Eligible Individuals in Environmentally Burdened Communities Through Enhanced Risk Communication
Brief Title: Project PLUS Lung Cancer Screening Promotion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Principal Investigator, Katharine Rendle, Assistant Professor, Abramson Cancer Center at Penn Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UPCC 03523; 849953 (Other: UPenn IRB)
Record Dates: First submitted 2023-06-29; First posted 2023-07-10 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2024-05

CONDITIONS: Lung Cancer
Keywords: Screening
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): This arm includes patients who view the integrated health video that provides information about both smoking and environmental risk.
  Interventions: Behavioral: Intervention video
- Control Video Arm (Experimental): This arm includes patients who view the integrated health video that provides information ONLY about smoking risk.
  Interventions: Behavioral: Control video

INTERVENTIONS:
Behavioral: Intervention video — This intervention is an integrated health video provides individual (smoking) and environmental risk communication on intention to obtain lung cancer screening.
  Arms: Intervention Arm
Behavioral: Control video — This intervention is an integrated health video provides individual (smoking) risk communication on intention to obtain lung cancer screening.
  Arms: Control Video Arm

SUMMARY:
Project PLUS is a pilot study that aims to develop and obtain preliminary feasibility and efficacy data on an enhanced risk communication approach to promote lung cancer screening (LCS) intentions among screening-eligible individuals from environmentally burdened communities. Project PLUS will combine qualitative interviews to explore subject awareness regarding lung cancer risk and air pollution, barriers to LCS, and perceptions regarding risk communication messaging, develop a health education video, and a between-subjects experiment to compare Data from this pilot will form the basis for enhanced community engagement efforts and subsequent communication research to examine the effectiveness of incorporating the involuntary air pollution risk information in risk communication interventions. The long term goal is to reduce lung cancer burden and disparities among environmentally burdened communities within and outside of Philadelphia.

DETAILED DESCRIPTION:
Project PLUS is a pilot study that aims to develop and obtain preliminary feasibility and efficacy data on an enhanced risk communication approach to promote lung cancer screening (LCS) intentions among screening-eligible individuals from environmentally burdened communities. Project PLUS will combine qualitative interviews to explore subject awareness regarding lung cancer risk and air pollution, barriers to LCS, and perceptions regarding risk communication messaging, develop a health education video, and a between-subjects experiment to compare Data from this pilot will form the basis for enhanced community engagement efforts and subsequent communication research to examine the effectiveness of incorporating the involuntary air pollution risk information in risk communication interventions. The long term goal is to reduce lung cancer burden and disparities among environmentally burdened communities within and outside of Philadelphia.

This study is guided by the Health Belief Model and the Reasoned Action Approach.1 The study team will engage with two community partner organizations (Chester Environmental Partnership and Clean Water Action) to obtain feedback in implementing the study procedures and input on content for the health education video. The long-term goal is to improve LCS and reduce racial, ethnic, and socioeconomic disparities in lung cancer mortality.

ELIGIBILITY:
Patient interview participants will be eligible if they:

1. Are ages 50 - 80 years;
2. Have a history of at least 20 cigarette pack-years, and who have quit within the past 15 years or are currently smoking;
3. Had a primary care visit at Penn Medicine within the last two years (2020-2021);
4. Have documented history of lung cancer screening or lung cancer
5. Are residing in one of 10 eligible zip codes;
6. Are English-speaking;
7. Are able to view the study videos;
8. Are able to participate in a video-conference interview using a HIPAA-compliant platform or able to participate in an interview over the phone.

Pilot trial participants will be eligible if they:

1. Are ages 50 - 80 years;
2. Are documented history of at least 20 cigarette pack-years, and who have quit within the past 15 years or are currently smoking;
3. Have no documented history of lung cancer screening or lung cancer;
4. Did not participate in patient interviews;
5. Had a primary care visit at Penn Medicine within the last two years (2020-2022);
6. Are residing in one of 10 eligible zip codes;
7. Are English-speaking;
8. Are able to view the study videos and complete an online survey.

Key Exclusion Criteria:

Patient interview participants are excluded if:

a. They are not eligible for lung cancer screening.

Pilot trial participants are excluded if they:

1. Do not meet inclusion criteria;
2. Participated in patient interviews.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
The number of patients who intend or do obtain lung cancer screening within the next 3 months. | Assessed immediately after viewing the health education video.
  This outcome will be measured using a post-test survey given to patients immediately after viewing a health education video assessing the patient's intention to obtain a lung cancer screening within the next 3 months.

SECONDARY OUTCOMES:
Completion of lung cancer screening | 6 months of study enrollment
  The study team will utilize chart review and medical record data to assess whether patients scheduled or received a lung cancer screening within 6 months of enrollment in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Katharine Rendle, PhD,MSW,MPH, Principal Investigator — University of Pennsylvania; Andy Tan, PhD,MPH,MBA, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No